CLINICAL TRIAL: NCT02832492
Title: Does Pupil Near Response Have Prognostic Value in Patients With Unresponsive Wakefulness Syndrome?
Brief Title: The Prognostic Value of Pupil Near Response in UWS Patients
Status: Completed | Type: Observational
Sponsor: Wentao Zeng (Other)
Responsible Party: Sponsor-Investigator, Wentao Zeng, Master degree candidate, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Other Study IDs: 2015/1030/B
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Vegetative State
Keywords: disorders of consciousness; unresponsive wakefulness syndrome; pupil near response; prognosis of consciousness recovery
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PNR+: Patients who will show pupil near response during PNR assessment.
  Interventions: Behavioral: pupil near response
- PNR-: Patients who will not show pupil near response during PNR assessment.
  Interventions: Behavioral: pupil near response

INTERVENTIONS:
Behavioral: pupil near response

SUMMARY:
Previous studies suggest that the stimulus of pupil near response (PNR) may be a conscious perception of a blurred image. Moreover, PNR is a reflex that can be objectively observed and with no motor output, suggesting it might be a more convenient index for consciousness evaluation and consciousness recovery in patients with disorders of consciousness (DOC). We thus hypothesized that PNR+ patients (patients show PNR during the assessment) would have better prognosis than PNR- patients (patients fail to show PNR during the assessment).Based on this hypotheis, researchers will assess pupil near response in patients with unresponsive wakefulness syndrome (UWS) and compare the prognosis difference between PNR+ patients and PNR- patients to assess its prognosis value.

DETAILED DESCRIPTION:
PNR assessments will be conducted in patients with Unresponsive Wakefulness Syndrome (UWS) diagnosed by the Coma recovery scale-revised (CRS-R).An objective index,the ratio of pupillary constriction (pupil diameter change after a stimulus presentation divided by the resting state pupil diameter) will be used as the measure of PNR's presence (positive results indicate the presence of PNR,whereas negative results indicate the absence of PNR).According to the presence of PNR,patients will be divided into 2 groups,one includes patients who show PNR during the PNR assessment (PNR+),the other includes patients who fail to show PNR during the PNR assessment(PNR-).3 months later,a follow-up will be conducted to obtain their prognosis in the form of another CRS-R assessment.Patients diagnosed as Minimally Conscious State (MCS) will be considered as favourable prognosis,patients diagnosed as UWS will be considered as unfavourable prognosis.Their prognosis difference will then be compared to see PNR's effect on their prognosis (consciousness recovery). And for they couldn't show conscious visual behaviors (visual behaviors in CRS-R which indicate MCS) in the first CRS-R,their difference between visual prognosis (difference between each group's proportion of patients showing conscious visual behavior diagnosed by CRS-R in the follow up) will be compared to see PNR's capability to predict prognosis in patients without voluntary eye movements (conscious visual behaviors in CRS-R require voluntary eye movements).

Researchers expect to see the PNR+ group have better prognosis in both comparison.

ELIGIBILITY:
Inclusion Criteria:

* unresponsive wakefulness syndrome (diagnosed by CRS-R)
* normal or corrected to normal vision before the incidence (myopia did not exceed 300 degrees Fahrenheit, farsightedness was less than + 2.00 d)
* positive pupil light reflex.

Exclusion Criteria:

* nystagmus and drooping eyelids
* unstable vital signs
* under sedation during PNR test.

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who has been diagnosed as unresponsive wakefulness syndrome by CRS-R before this study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

PRIMARY OUTCOMES:
Each group's proportion of MCS patients diagnosed by CRS-R in the follow up | 3 months after pupil near response assessment in this study
  Greater proportion in PNR+ group suggests PNR has prognostic value to DOC patients thus has relationship with consciousness

SECONDARY OUTCOMES:
Each group's proportion of recovery of conscious visual function diagnosed by visual subscale of CRS-R in the follow up | 3 months after pupil near response assessment in this study
  Greater proportion in PNR+ group suggests PNR can correct misdiagnosis caused by lesions on motor systems thus is applicable to patients without motor function